CLINICAL TRIAL: NCT03632005
Title: A Prospective Randomized Clinical Trial Comparing Incisional Negative Pressure Wound Therapy to Conventional Sterile Dressing in Patients Undergoing Thoracolumbar Posterior Spine Surgery
Brief Title: Negative Pressure Wound Therapy vs. Sterile Dressing for Patients Undergoing Thoracolumbar Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: John Street (Other)
Collaborators: KCI USA, Inc (Industry); University of British Columbia Orthopaedics Research Excellence Fund (Unknown)
Responsible Party: Sponsor-Investigator, John Street, Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H13-02263
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Disease; Spinal Cord Injury; Spinal Degeneration; Spinal Deformity
Keywords: Surgical Site Infection
MeSH Terms: conditions — Neoplasm Metastasis; Spinal Cord Injuries; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sterile Dressing (Other): Standard of care treatment - Standard wound care involves the application of an occlusive dressing in the operating room, a dressing change on Post-operative Day 3 and then dressing changes as needed until suture/staple removal on Post-operative Day 14.
  Interventions: Other: Sterile dressing
- Vacuum Assisted Closure (Active Comparator): The Prevena™ System, a type of vacuum assisted closure, is indicated for use over clean, closed incisions that continue to drain following sutured or stapled closure. It acts by removing exudate, helping hold the edges of the incision together, protecting the surgical site from external contamination in a clean, protected postoperative wound environment.
  Interventions: Device: Vacuum Assisted Closure

INTERVENTIONS:
Device: Vacuum Assisted Closure — Patients will be randomized to receive either standard dressing changes or the Prevena™ System on the day of their operation.
  Other Names: Prevena™ System
  Arms: Vacuum Assisted Closure
Other: Sterile dressing — Standard wound care involves the application of an occlusive dressing in the operating room, a dressing change on Post-operative Day 3 and then dressing changes as needed until suture/staple removal on Post-operative Day 14.
  Arms: Sterile Dressing

SUMMARY:
The purpose of this study is to determine if the use of the Prevena™ System decreases the rate of subcutaneous seroma, superficial wound dehiscence and infection.

DETAILED DESCRIPTION:
Certain risk factors have been identified in patients that may lead to poor wound healing or infection. Many things have been tried to decrease this risk (more antibiotics, different types of stitches, etc) but very few have been shown to be of any significant benefit.

The use of a special vacuum dressing called the Prevena™ System, which has received approval from Health Canada for the management of closed surgical incisions, has been shown to be of some benefit in hip surgery where wounds are identified as being "at risk." Vacuum dressings have been used with great success in patients with open wounds and have resulted in fewer infections and wound related complications. It is thought that if vacuum dressings can be used in the treatment of existing wounds, then maybe they can be used preventatively before there is a problem with the wound.

Standard wound care after spine surgery involves a dressing that seals the wound for 72 hours after surgery and is then changed on a daily basis until the surgical sutures or staples are ready to be removed. This has been routine for many years.

The purpose of this study is to see if using a vacuum dressing (Prevena™ System) will decrease the number of infections and/or clinic and hospital visits for wound related issues compared to using a standard dressing on wounds in patients with risk factors for early wound infection.

ELIGIBILITY:
Inclusion Criteria: Patients who meet the following criteria are eligible for admission into the study:

* Require spine surgery with a posterior midline incision that involves the thoracic, lumbar and/or sacral spine
* Capable of and agree to consent and randomization
* Be in one of the following clinical presentation groups:

  1. Metastic tumor of the thoracic or lumbar spine (T1-S5), requiring instrumentation and decompression, with or without pre-operative radiation to surgical site
  2. Thoracolumbar degeneration or deformity (T1-S5) with index surgery >6 months prior, requiring revision surgery with additional instrumentation
  3. Acute traumatic thoracolumbar (T1-L5) fracture(s) with neurological deficit (AIS A-C), requiring instrumentation and decompression

All study participants will remain in hospital for a minimum of 7 days post-op as per standard of care. As a result, the full duration of application of the Prevena dressing will take place in hospital.

Exclusion Criteria: patients who fulfill any of the following criteria are not eligible for admission into the study:

* Undergoing percutaneous surgery
* Active Surgical Site Infection (SSI) or primary spinal column infection or distant site infection (urinary tract, respiratory tract, etc.) at time of admission
* Pregnancy

The following are clinical scenarios that would mandate the patients' exclusion from final analysis:

* Failure to complete the 6-week clinical follow-up (Lost to Follow Up)
* Second surgery required, at the same anatomical site, during study time period (six weeks), for causes other than primary (SSI) or secondary (dehiscence, seroma) study endpoints

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2017-03-18 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute, post-operative surgical site infection (SSI) following thoracolumbar spinal surgery for a metastatic tumor, revision requiring additional instrumentation or acute traumatic spinal cord injury | 6 weeks post-op
  Based on visual inspection of the surgical site, a 'Wound Inspection & Dressing Utilization' case report form will be completed by a clinician, concluding at Week 6 post-op, to assess for the presence of SSI.

CONTACTS AND LOCATIONS:
Overall Officials: John Street, MD,PhD,FRCSI, Principal Investigator — University of British Columbia & Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No